CLINICAL TRIAL: NCT02380066
Title: Proof Of Concept Study of Anyu Peibo in the Treatment of Major Depressive Disorder(MDD): a Randomized, Double-Blind, Placebo-Paralleled,Dose-Finding, Multicenter Clinical Trial
Brief Title: Comparison of Anyu Peibo With Placebo in Treatment of MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Su Zhou YiHua Biotechnology Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYPB-MDD-Ⅱa-1401; 2012ZX09303-003 (Other Grant/Funding Number: China National Major Project)
Record Dates: First submitted 2015-02-13; First posted 2015-03-05 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2015-03

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Anyu Peibo 0.4g per day (Experimental): Anyu Peibo Capsule, oral, 0.2g twice per day
  Interventions: Drug: Anyu Peibo
- Anyu Peibo 0.8g per day (Experimental): Anyu Peibo Capsule, oral, 0.4g twice per day
  Interventions: Drug: Anyu Peibo
- Anyu Peibo 1.2g per day (Experimental): Anyu Peibo Capsule, oral, 0.6g twice per day
  Interventions: Drug: Anyu Peibo
- Anyu Peibo 1.6g per day (Experimental): Anyu Peibo Capsule, oral, 0.8g twice per day
  Interventions: Drug: Anyu Peibo
- Placebo (Placebo Comparator): Placebo,oral, twice per day
  Interventions: Drug: Anyu Peibo

INTERVENTIONS:
Drug: Anyu Peibo — Placebo
  Other Names: Placebo

SUMMARY:
The purpose of this study is to determine whether Anyu Peibo Capsule in different doses are effective in the treatment of Depression.

And to explore the preliminary information of safety and efficacy of Anyu Peibo Capsule in the Chinese Patients with Depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult with primary diagnosis of major depressive disorder(MDD) based on the criteria of DSM-IV-TR, single episode or recurrent episode, not accompanied with psychotic symptoms. Coding of diagnosis included: 296.21 MDD single episode, mild 296.22 MDD single episode, moderate 296.31 MDD recurrent episode, mild 296.32 MDD recurrent episode, moderate
* The total score of HAMD-17 is ≥18 and ≤24 in both screening visit and baseline visit.
* The subject understands and consents to takes part in this clinical trials. The subjects should sign informed consent.

Exclusion Criteria:

* The subject has a significant risk of suicide according to the investigator's opinion or has a score ≥3 on item 3(suicide assessment) of the HAMD or has made a suicide attempt.
* The subject has a current DSM-Ⅳ-TR axisⅠpsychiatric diagnosis other than depression.
* When the HAMD17 score of baseline visit compares with the screening visit, the decreasing rate is ≥25%.
* Any unstable cardiovascular, hepatic, renal, endocrine(thyroid gland dysfunction), blood,or other medical disease.
* Had a history of seizure disorder,except infantile febrile convulsion.
* The subject has accepted psychosurgery or electroconvulsive therapy within 3months.
* With psychotic symptoms.
* The subject has a history of mania episode, including manic, mixed or rapid cycle attack.
* The subject has a current diagnosis or history of depression due to any other psychotic disorder or a general medical condition.
* The subject with refractory depressive disorder,i.e.the patients who used at least two different mechanisms antidepressants with adequate dosage and duration treatment still had no respond.
* Clinically significant electrocardiographic(ECG) abnormalities or abnormal laboratory values(eg. Hepatic function above 1.5 times of clinical toplimit, renal function or thyroid gland function index above toplimit, routine blood, fasting blood glucose value above or below 1.1 times of the upper limit of normal or in 1.1 times with the clinical significance of abnormality).
* The subject has a diagnosis of alcohol or other substance abuse or dependence at least 1 years prior to the baseline visit.
* Known hypersensitivity to Big Leaf Ju, or at least to two kinds of drugs, or serious allergic physique.
* Women who were pregnant, breast-feeding, or planning to become pregnant during study. Men who have request to fertility during study period. The subject could not take safe and effective birth control measures.
* The subject could not take medication according to the doctor's advice. i.e. the compliance of the subject is poor.
* The subject uses antidepressant drug normally before 2 weeks of screening, and stops using psychotropic drug less than 7 half-life period (monoamine oxidase inhibitor more than 2 weeks, fluoxetine more than 1 month).
* The subject has participated in a drug clinical trial within 1 month before screening.
* The investigator think the subject is unsuitable to enrol in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The change of total score from baseline in MADRS scale | 6 weeks

SECONDARY OUTCOMES:
clinical response rate according to MADRS | 6 weeks
clinical remission rate according to MADRS | 6 weeks
CGI(CGI-S,CGI-I) | 6 weeks
The change of total score from baseline in HAMD scale | 6 weeks
decreasing rate from baseline in HAMD scale | 6 weeks
clinical response rate according to HAMD | 6 weeks
clinical remission rate according to HAMD | 6 weeks
change from baseline in HAMA | 6 weeks

OTHER OUTCOMES:
vital sign | 6 weeks
  Blood pressure, heart rate, temperature and respiratory rate
AE(adverse events) | 6 weeks
laboratory examination | 6 weeks
  Blood RT, Urinalysis,Hepatic function,Renal function,FBG,Lipid,CK,HBV,Thyroid Function Test and U-HCG
ECG | 6 weeks
C-SSRS | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD PhD, Principal Investigator — Shanghai Mental Health Center
Locations (6):
- China (6):
  - Anhui province hospital of TCM, Hefei, Anhui
  - Guang'anmen Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Guangzhou Huiai Hospital, Guangzhou, Guangdong
  - Jiangsu province hospital of TCM, Nanjing, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu